CLINICAL TRIAL: NCT02724046
Title: Cluster-randomized Trial to Evaluate the Impact of Ciprofloxacin for Contacts of Cases of Meningococcal Meningitis as an Epidemic Response
Brief Title: Ciprofloxacin for the Prevention of Meningococcal Meningitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Epicentre (Other)
Collaborators: Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Ciprofloxacin chemoprophylaxis
Record Dates: First submitted 2016-03-15; First posted 2016-03-31 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Meningitis, Meningococcal
Keywords: Neisseria meningitidis; Ciprofloxacin; Chemoprevention
MeSH Terms: conditions — Meningitis, Meningococcal | interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard care (No Intervention): No chemoprevention for contacts of cases of meningitis (current standard of care) with a health promotion visit by a study nurse after the first notification of cases during the epidemic
- Household prophylaxis (Active Comparator): Chemoprophylaxis with a single dose of oral ciprofloxacin for household members of reported cases of meningitis. For participants age >12 years: 500 mg tablet; age 5-12 years: 250 mg tablet; age 1-4 years: 125 mg tablet; age 3-11 months: 100 mg (2 ml oral suspension); age <3 months: 75 mg (1.5 ml oral suspension).
  Interventions: Drug: Ciprofloxacin
- Village prophylaxis (Active Comparator): Chemoprophylaxis with ciprofloxacin in the setting of a village-wide distribution after the notification of the first case of meningitis in a village. For participants age >12 years: 500 mg tablet; age 5-12 years: 250 mg tablet; age 1-4 years: 125 mg tablet; age 3-11 months: 100 mg (2 ml oral suspension); age <3 months: 75 mg (1.5 ml oral suspension).
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: Ciprofloxacin — Single-dose oral ciprofloxacin
  Other Names: Cipro
  Arms: Household prophylaxis; Village prophylaxis

SUMMARY:
This study evaluates the effect of antibiotic prophylaxis with ciprofloxacin, given to the contacts of meningitis cases, on the overall attack rate of meningitis during an epidemic. One third of enrolled villages will receive standard care; in one-third of villages, household contacts of meningitis cases will be offered a single dose of oral ciprofloxacin; and in one-third of villages, the entire village will be offered a single dose of oral ciprofloxacin after the notification of the first case in the village.

DETAILED DESCRIPTION:
Antibiotic prophylaxis is not currently recommended for contacts of cases during a meningitis epidemic in the African Meningitis Belt. Reactive vaccination campaigns are the preferred strategy for prevention during an epidemic.

A novel strain of meningococcus, Neisseria meningitidis serogroup C (NmC), began circulating in Nigeria in 2013 and caused a major epidemic with over 10 000 cases in Nigeria and Niger in 2015.

There is currently a global shortage of vaccine against NmC, and a recent WHO expert panel called for the formal evaluation of antibiotic prophylaxis as another epidemic response strategy.

When taken as a single dose, oral ciprofloxacin effectively eliminates nasopharyngeal carriage of meningococcus.

This trial aims to investigate two different antibiotic prophylaxis strategies during an epidemic of meningococcal meningitis: ciprofloxacin prophylaxis to household members of cases and village-wide prophylaxis after the notification of a case in a village. These two strategies will be compared to villages receiving standard care.

ELIGIBILITY:
Inclusion Criteria:

* Resident in a village included in the study area

Exclusion Criteria:

* Patients currently exhibiting symptoms of meningitis (to be immediately referred for further care)
* Persons with a known allergy to fluoroquinolone antibiotics.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-04-22 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-06-12 (Actual)

PRIMARY OUTCOMES:
Meningitis Attack Rate | From enrollment of a village through study completion, an average of 3 months
  The primary outcome aims to evaluate the impact of a chemoprevention strategy as a public health intervention during a meningitis outbreak, which is best evaluated by looking at the overall attack rates in the study area.

SECONDARY OUTCOMES:
Proportion of participants with ciprofloxacin-resistant enterobacteriaceae in their stools | Prior to ciprofloxacin dosing (day 0) and at 7 days and 28 days post-ciprofloxacin dosing
  A substudy is proposed to compare rates of acquisition of ciprofloxacin resistance among participants in the standard care arm and participants in the village prophylaxis arm. 20 participants in 10 villages in each of the two arms will be asked to provide stool samples on days 0, 7 and 28
Proportion of patients who received ciprofloxacin who develop meningitis | From enrollment of a village through study completion, an average of 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca F Grais, PhD, Study Director — Epicentre
Locations (1):
- Madarounfa Health District, Madarounfa, Maradi Region, Niger

IPD SHARING:
Plan to Share IPD: Yes
A de-identified data set can be made available after the signature of an appropriate data sharing agreement.

REFERENCES:
- [Derived] Coldiron ME, Assao B, Page AL, Hitchings MDT, Alcoba G, Ciglenecki I, Langendorf C, Mambula C, Adehossi E, Sidikou F, Tassiou EI, De Lastours V, Grais RF. Single-dose oral ciprofloxacin prophylaxis as a response to a meningococcal meningitis epidemic in the African meningitis belt: A 3-arm, open-label, cluster-randomized trial. PLoS Med. 2018 Jun 26;15(6):e1002593. doi: 10.1371/journal.pmed.1002593. eCollection 2018 Jun. PMID 29944651
- [Derived] Coldiron ME, Alcoba G, Ciglenecki I, Hitchings M, Djibo A, Page AL, Langendorf C, Grais RF. Ciprofloxacin for contacts of cases of meningococcal meningitis as an epidemic response: study protocol for a cluster-randomized trial. Trials. 2017 Jun 24;18(1):294. doi: 10.1186/s13063-017-2028-y. PMID 28646924